CLINICAL TRIAL: NCT01068470
Title: Lymphokine Activated Killer (LAK) Cell Activity Against Cell Lines In-vitro of LAK Generated in Vivo by Pulse Interleukin-2 Therapy
Brief Title: Determining the Lymphokine Activated Killer (LAK) Cytotoxicity Present in Patients Undergoing Interleukin-2 Therapy
Acronym: LAK
Status: Terminated | Type: Observational
Why Stopped: PI left the institution
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 59210
Record Dates: First submitted 2010-02-11; First posted 2010-02-15 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Melanoma; Kidney Cancer
Keywords: Interleukin-2; Melanoma; Kidney Cancer; Lymphokine Activated Killer cells
MeSH Terms: conditions — Melanoma; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with melanoma or kidney cancer

SUMMARY:
Therapy with Interleukin-2 stimulates lymphocytes in humans to become Lymphokine-activated Killer cells (LAK). This study will determine if these killer cells are able to kill certain standard cell-lines in the laboratory.

DETAILED DESCRIPTION:
Blood samples will be taken from patients undergoing outpatient Interleukin-2 therapy to measure the LAK cytotoxicity at baseline, after 1 cycle of therapy and 2 months later. The LAK cytotoxicity assay will be a standard colorimetric assay that measures lactic dehydrogenase release from lysed cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be undergoing Interleukin-2 therapy under the care of physicians at Loma Linda University Cancer Center
* Patients must sign and give written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Patients not undergoing Interleukin-2 therapy under the care of physicians at Loma Linda University Cancer Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Interleukin-2 therapy under the care of physicians at Loma Linda University Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
LAK cytotoxicity | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Walter Quan, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Cancer Center, Beaumont, California, United States